CLINICAL TRIAL: NCT03815188
Title: Use of the SonoSite Probe for Measuring Jugular Venous Pressure
Acronym: PRAGUE
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Other Study IDs: STH20529
Record Dates: First submitted 2019-01-21; First posted 2019-01-24 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-08

CONDITIONS: Aortic Valve Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Heart Valve Surgery: Pre-operative patients undergoing heart valve surgery will be selected and data recorded from each patient on the day of their surgery. This patient cohort is required in order to be able to accurately measure their JVP upon physical examination. Patients must have a central line inserted as part of their ongoing clinical management.

SUMMARY:
This prospective study will be performed in the Cardiothoracic (Chesterman) Department at Sheffield Teaching Hospitals NHSFT, Northern General Hospital. Pre-operative patients undergoing surgical valvular intervention, breathing both spontaneously and mechanically will be included in the trial. All patients will already have a central venous catheter inserted as part of their ongoing care. Patients will be eligible for the study irrespective of diagnosis or neck size. Patient demographical data will be recorded by Sam Jenkins following written consent, the day before the trial.

The goal of this study is to determine if ultrasound assessment of Jugular Venous Pressure (JVP) accurately predicts Central Venous Pressure (CVP). Secondary objectives aim to identify if using the angle of Louis to approximate the location of the right atrium produces inaccuracies when measuring JVP. Comparing results in patients breathing spontaneously or under positive pressure ventilation will identify if the form of ventilation impacts on JVP and CVP recording. Correlating results between physical JVP examination and ultrasound assessment of JVP to measure CVP will conclude if ultrasound is a more appropriate tool, in an era where the physical examination of the cardiovascular system is becoming less valuable.

DETAILED DESCRIPTION:
Initial exploratory investigations will compare left-sided and right-sided Jugular Venous Pressure (JVP) using ultrasonography. Should results show that they are the same, the central line is to be placed into the right internal jugular vein when required.

To begin the trial and whilst the patient is spontaneously breathing, a physical examination of the right JVP will be performed. A central line will be inserted with the patient awake into the right internal jugular vein. Left-sided ultrasound of JVP and Central Venous Pressure (CVP) will be measured using the right-sided catheter will be recorded simultaneously. The tip of the catheter attached to the transducer (which is zeroed to the reference point) will be placed at the point of venous collapse, identified by ultrasonography, to identify if the JVP and CVP match. The tip of the catheter will then be placed at the angle of Louis. Measurement of the pressure difference between the angle of Louis and the reference point will identify if this value shows variability compared to previous approximations of 5cm above the right atrium. With the patient anaesthetised and mechanically breathing, left JVP and CVP will be measured once more. Twenty-four hours post-surgery, ultrasound of the JVP and CVP will be measured with the patient breathing spontaneously.

The physical JVP examination will be recorded from the opposite side to the central venous catheter. The bed will be adjusted to an angle between 30 and 60 degrees, that most clearly identifies the collapsing vein. Differentiation between the JVP and the carotid pulse must be distinguished. Tangential lighting using a flashlight should be used to correctly identify and note the apex of the jugular venous pulsations. Recordings will be taken at end-expiration allowing the vertical distance between the venous meniscus and phlebostatic axis to be measured. JVP will be measured in millimetres of water.

Ultrasound recordings will be made using the SonoSite ultrasound probe by Sam Jenkins. The equipment and gels required are used routinely on site and will be supplied by Sheffield Teaching Hospitals. The SonoSite probe will be calibrated prior to each use, based on the recommendations of the manufacturer. The angle of the bed is kept constant and the patient will remain in the same position following the physical JVP examination. Ultrasound gel will be applied, again on the opposite side to the central venous catheter. Locating the area of venous collapse will be identified following visualisation from both longitudinal and transverse planes. The apex of venous collapse at end-expiration will be marked using the longitudinal view. Corroboration of the correct position of the probe by looking at the transverse view will be performed prior to marking of venous collapse.

CVP will be measured once the central venous catheter has been zeroed. The reference point of the transducer will be placed at the 4th intercostal space, mid-axillary line. The bed should still be kept at a constant angle for this measurement. The mean of the 'a' wave upon end-expiration will be taken. Converting the CVP from millimetres of mercury to millimetres of water will allow direct comparison to prior findings of JVP.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery
* Patients who have a central line inserted during surgery
* Patients able and willing to give consent in verbal and written English.

Exclusion Criteria:

* Patients under the age of 18
* Patients unable to provide consent in verbal and written English
* Patients with thyroid enlargement or alternative reason causing obstruction to venous anatomy
* Patients with significant tricuspid regurgitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pre-operative patients undergoing heart valve surgery will be selected and data recorded from each patient on the day of their surgery. This patient cohort is required in order to be able to accurately measure their JVP upon physical examination. Patients must have a central line inserted as part of their ongoing clinical management. Patients will be selected based on the weekly surgery schedule and will require participation of the anaesthetist. The anaesthetist will be required to insert the central line, anaesthetise the patient and adjust the transducer when asked.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Ultrasonography | Through study completion - 30/09/2019
  Ultrasonography is expected to be a more accurate measure of CVP compared to physical JVP examination and is hypothesised to accurately predict CVP.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Teaching Hospitals NHS FT, Sheffield, England, United Kingdom

REFERENCES:
- [Background] Brennan JM, Blair JE, Goonewardena S, Ronan A, Shah D, Vasaiwala S, Brooks E, Levy A, Kirkpatrick JN, Spencer KT. A comparison by medicine residents of physical examination versus hand-carried ultrasound for estimation of right atrial pressure. Am J Cardiol. 2007 Jun 1;99(11):1614-6. doi: 10.1016/j.amjcard.2007.01.037. Epub 2007 Apr 18. PMID 17531592
- [Background] Cook DJ, Simel DL. The Rational Clinical Examination. Does this patient have abnormal central venous pressure? JAMA. 1996 Feb 28;275(8):630-4. No abstract available. PMID 8594245
- [Background] Deol GR, Collett N, Ashby A, Schmidt GA. Ultrasound accurately reflects the jugular venous examination but underestimates central venous pressure. Chest. 2011 Jan;139(1):95-100. doi: 10.1378/chest.10-1301. Epub 2010 Aug 26. PMID 20798190
- [Background] Fletcher RH, Fletcher SW. Has medicine outgrown physical diagnosis? Ann Intern Med. 1992 Nov 1;117(9):786-7. doi: 10.7326/0003-4819-117-9-786. No abstract available. PMID 1416582
- [Background] Jang T, Aubin C, Naunheim R, Char D. Ultrasonography of the internal jugular vein in patients with dyspnea without jugular venous distention on physical examination. Ann Emerg Med. 2004 Aug;44(2):160-8. doi: 10.1016/j.annemergmed.2004.03.014. PMID 15278091
- [Background] Lipton B. Estimation of central venous pressure by ultrasound of the internal jugular vein. Am J Emerg Med. 2000 Jul;18(4):432-4. doi: 10.1053/ajem.2000.7335. PMID 10919533
- [Background] Mangione S, Nieman LZ. Cardiac auscultatory skills of internal medicine and family practice trainees. A comparison of diagnostic proficiency. JAMA. 1997 Sep 3;278(9):717-22. PMID 9286830
- [Background] Seth R, Magner P, Matzinger F, van Walraven C. How far is the sternal angle from the mid-right atrium? J Gen Intern Med. 2002 Nov;17(11):852-6. doi: 10.1046/j.1525-1497.2002.20101.x. PMID 12406357
- [Background] Socransky SJ, Wiss R, Robins R, Anawati A, Roy MA, Yeung IC. Defining normal jugular venous pressure with ultrasonography. CJEM. 2010 Jul;12(4):320-4. doi: 10.1017/s1481803500012409. PMID 20650024
- [Background] Sondergaard S, Parkin G, Aneman A. Central venous pressure: we need to bring clinical use into physiological context. Acta Anaesthesiol Scand. 2015 May;59(5):552-60. doi: 10.1111/aas.12490. Epub 2015 Feb 13. PMID 25684176
- [Derived] Jenkins S, Knowles P, Briffa N. Portable ultrasound assessment of jugular venous pressure is an accurate method for estimating volaemic status in patients with cardiac disease. J Ultrasound. 2022 Dec;25(4):939-947. doi: 10.1007/s40477-022-00654-7. Epub 2022 Mar 15. PMID 35292924